CLINICAL TRIAL: NCT04220671
Title: Health Effects of Utilising Curative Health System Contacts to Provide Measles Vaccination - a Randomised Controlled Trial
Brief Title: Measles Vaccination at Health System Contacts
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 053/CNES/INASA/2019
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Measles Vaccine; Hospital Admission; Mortality; Non-specific (Heterologous) Effects of Vaccines
MeSH Terms: interventions — Measles Vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Standard dose measles vaccine, 0.5 ml
  Interventions: Biological: measles vaccine
- Control (Placebo Comparator): Saline injection, 0.5 ml
  Interventions: Other: Saline

INTERVENTIONS:
Biological: measles vaccine — Measles vaccine, Edmonston-Zagreb strain, 0.5 ml administered as a subcutaneous injection
  Arms: Intervention
Other: Saline — 0.9% NaCl
  Arms: Control

SUMMARY:
In addition to protecting against measles infection, measles vaccine (MV) strengthens the individual's ability to combat infections in general - MV has beneficial non-specific effects (NSE) lowering the risk of death and admissions by around 30%.

In Guinea-Bissau 30% of children do not receive a routine MV scheduled at 9 months of age, putting both the individual child's health and measles eradication at risk. The coverage of a second dose of MV, which was added to the Bissau-Guinean vaccination programme in 2022, is even lower. WHO recommends vaccination at health system contacts, including those for curative services. At the paediatric ward of the national hospital in Guinea-Bissau, there are more than 2600 yearly contacts with measles-un or under-vaccinated children aged 9-59 months, but no vaccines are given. In a randomised controlled trial, we will assess the effect of providing MV vs placebo to 5400 children at hospital contacts (at discharge or after an out-patient consultation) to test the hypothesis that MV reduces the risk of admission or death (composite outcome) by 25% over the subsequent 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Measles-unvaccinated children
* 9-59 months with a hospital contact (discharged or outpatient consultation) at the paediatric ward at the national hospital Simao Mendes.

Measles-under-vaccinated children (received first but not second dose of MV)

* 15-59 months with a hospital contact (discharged or outpatient consultation) at the paediatric ward at the national hospital Simao Mendes.

Exclusion Criteria:

* Axil temperature >38.0
* Mid upper arm circumference <110 mm

Ages: 9 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5400 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Non-accident mortality or admission (Composite outcome) | 6 months
  Composite outcome of non-accidental death (recorded through telephone interviews and passive case detection) or an identified non-accidental hospital admission at the national hospital Simao Mendes

SECONDARY OUTCOMES:
Non-accidental mortality | 6 and 12 months
  Non-accidental mortality. For the secondary outcomes, censoring will be applied for children whom we do not succeed to contact by telephone
Non-accidental hospital admission with an overnight stay in any health facility | 6 months
  Since we rely on passive case detection at the national hospital, we will not censor analysis time of children with no information by telephone interviews in the primary analysis. For the secondary outcomes, censoring will be applied for children whom we do not succeed to contact by telephone
Cause specific hospital admissions at the national hospital. | 6 months
  classifying admissions in the main categories: Respiratory infections, Gastro-intestinal infections, Sepsis, Malaria and other

OTHER OUTCOMES:
Adverse events | 2 weeks
  Registered contacts with the health system (information on consultations or admissions during the first 2 weeks after enrolment identified through the registration system at the national hospital and registration of outpatient consultations at the health centres in the study area. Among the first 1000 enrolled measles unvaccinated children: Home visits to assess specific symptoms and minor morbidity at day 2, 4, 7 and 14. Among the first 500 enrolled children who have received the first but not the second dose of MV: Telephone follow up after 7 and 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ane Fisker, MD, PhD, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: No
Provided request, data can be made available

REFERENCES:
- [Derived] Fisker AB, Martins JSD, Jensen AM, Martins C, Aaby P, Thysen SM. Health effects of utilising hospital contacts to provide measles vaccination to children 9-59 months-a randomised controlled trial in Guinea-Bissau. Trials. 2022 Apr 23;23(1):349. doi: 10.1186/s13063-022-06291-z. PMID 35461287